CLINICAL TRIAL: NCT01895400
Title: A Single-center, Prospective, Randomized, Parallel Group, Placebo-controlled Exploratory Study on the Effect of Renexin Tablet in Patients With Recurrent Vestibulopathy
Brief Title: Effect of Renexin Tablet in Patients With Recurrent Vestibulopathy
Acronym: REREV
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Participant enrollment is much delayed. The whole design needs to be revised.
Sponsor: Jong Woo Chung (Other)
Collaborators: SK Chemicals Co., Ltd. (Industry); Asan Medical Center (Other)
Responsible Party: Sponsor-Investigator, Jong Woo Chung, MD, Asan Medical Center
Organization: Asan Medical Center (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: AMC-2013-0165; 20130055275 (Other: KFDA)
Record Dates: First submitted 2013-07-05; First posted 2013-07-10 (Estimated); Last update posted 2016-02-17 (Estimated); Status verified 2016-02

CONDITIONS: Recurrent Vestibulopathy
Keywords: Renexin for Recurrent Vestibulopathy
MeSH Terms: conditions — Vestibular Neuronitis | interventions — renexin; Cilostazol; Ginkgo Extract

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Renexin (Active Comparator): Renexin 1T bid for 12 weeks
  Interventions: Drug: Renexin (cilostazol 100mg + gingko biloba extract 80 mg)
- Placebo (Placebo Comparator): Placebo 1T bid for 12 weeks
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Renexin (cilostazol 100mg + gingko biloba extract 80 mg) — Take Renexin 1T bid po medication for 8 weeks
  Other Names: Renexin
  Arms: Renexin
Drug: Placebo — Take placebo drug 1T bid po medication for 8 weeks
  Other Names: Renexin
  Arms: Placebo

SUMMARY:
The purpose of this study is to determine whether Renexin is effective in the treatment of vestibular symptoms in patients with recurrent vestibulopathy.

DETAILED DESCRIPTION:
1. Study design

   * Among patients who visitied for recurrent vertigo more than 3 months, patients will be included after ruling out other peripheral vertigo through history taking, physical examination, Dix-Hallpike test, head-thrust test.
   * Included patients will go through permission, laboratory tests (CBC, chemical battery, coagulation battery, urine HCG (only women of childbearing age), posturography. During patients selection period for inclusion(2 weeks), taking medication for vertigo is prohibited.
   * Included patients will be randomized to Treatment group (Renexin) and Placebo group.
   * All patients before treatment will do dizziness handicap inventory(DHI), visual analogue scale (VAS) for vertigo, questionnaire for quality of life (SF36).
   * After 4 weeks(+-~ 3 days) of drug administration, DHI, VAS for vertigo, SF36 will be done for drug compliance and side effects.
   * After 8 weeks(+-~ 3 days) of drug administration, posturography, DHI, VAS for vertigo, SF36 will be done for drug compliance and side effects.
   * For control of severe vertigo during drug administration, Valium 2mg can be used as a salvage treatment, and number of valium administration will be checked at every visit.
2. Statistical analysis

   * As a statistical analysis, paired T-test will be used to compare equilibrium score, DHI, VAS, SF-36. When p-value is <0.05, it will be considered as significant difference.

ELIGIBILITY:
Inclusion Criteria:

* Recurrent vestibulopathy patient with symptoms more than 3 months of recurrent vertigo
* Visual analogue scale (VAS) score between 4 to 8

Exclusion Criteria:

* Showing signs of central lesion in MRI or neurologic exams
* central nystagmus or loss of consciousness with vertigo
* cerebellar symptoms such as ataxia, dysarthria, gait disturbance
* Diagnosed as peripheral vertigo such as benign paroxysmal positional vertigo, Meniere's disease, migrainous vertigo in recent 3 months
* Bilateral vestibular dysfunction
* Vestibular neuronitis symptom appeared in recent 6 months
* Chronic liver disease (ALT>100 or AST>100) or chronic kidney disease (Creatinine > 3.0 mg)
* Blood Hemoglobin < 10mg/dl (in male) or < 8 mg/dl (in female)
* Contraindication for testing drug (ex. Pregnancy or breast feeding etc.)
* Taking antiepileptics such as phenobarbital, phenytoin, carbamazepine or rifampin in recent 2 weeks
* Taking cilostazol, gingko biloba for other disease
* Allergy/hypersensitivity to Renexin
* Severe drug toxicity when taking Renexin previously

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2013-07; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
equilibrium score of dynamic posturography | after 8 weeks of treatment
  compared with pretreatment equilibrium score

SECONDARY OUTCOMES:
dizziness handicap inventory | at 4 weeks, 8 weeks after treatment
  compared with pretreatment DHI score
visual analogue scale (VAS) of vertigo | at 4 weeks, 8 weeks after treatment
  compared with pretreatment VAS score
Questionnaire for Quality of life (SF36) | at 4 weeks, 8 weeks after treatment
  compared with pretreatment SF36 score

CONTACTS AND LOCATIONS:
Overall Officials: Jong Woo Chung, MD, Study Chair — Asan Medical Center
Locations (1):
- Asan Medical Center, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: Undecided
This study is decided to be terminated. Among 26 participants, 15 finished medication according to the protocol. I am not sure that these data can be analyzed because data is still unblinded.